CLINICAL TRIAL: NCT01376089
Title: A Phase 4 Randomized, Double-blind Study Comparing Patient Comfort and Safety Between Iodixanol 320 mg I/mL and Iopamidol 370 mg I/mL in Patients Undergoing Contrast-Enhanced Computed Tomographic (CECT) Imaging of the Abdomen/Pelvis
Brief Title: Iodixanol Versus Iopamidol in Patients Undergoing Contrast-Enhanced Computed Tomographic Imaging of Abdomen/Pelvis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GE-012-097
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-11

CONDITIONS: Patient Comfort and Safety
Keywords: Safety
MeSH Terms: interventions — iodixanol; Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1-Iodixanol (Other)
  Interventions: Drug: Iodixanol
- Arm 2-Iopamidol (Active Comparator)
  Interventions: Drug: Iopamidol

INTERVENTIONS:
Drug: Iodixanol — Iodixanol 320 mg I/mL as a single iv. administration.
  Other Names: Visipaque
  Arms: Arm 1-Iodixanol
Drug: Iopamidol — Comparator agent iopamidol (Isovue) 370 mg I/mL as a single iv. administration.
  Other Names: Isovue
  Arms: Arm 2-Iopamidol

SUMMARY:
The purpose of this study is to evaluate and compare overall patient comfort profile between the Iso-osmolar contrast media (IOCM), iodixanol 320 mg I/mL, and a Low-osmolar contrast media (LOCM), iopamidol 370 mg I/mL in patients undergoing Contrast-Enhanced Computed Tomographic (CECT) imaging of the abdomen/pelvis.

ELIGIBILITY:
Inclusion Criteria:

* The subject is over 18 years old.
* Subjects are referred to undergo a CECT imaging of the abdomen/pelvis as part of their routine clinical care.

Exclusion Criteria:

* The subject has known allergies to iodine or any prior history of adverse reaction to iodinated CM.
* The subject received another administration of CM within 24 hours prior to baseline or is scheduled to receive one within the 24 hour follow-up period.
* The subject is pregnant.
* The subject is taking metformin (e.g., Glucophage®) but is not willing or unable to discontinue at the time of the study procedure.
* The subject manifests thyrotoxicosis or is on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Lim, PharmD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 304 subjects were enrolled in this study, however, 5 subjects did not receive contrast media due to administrative and /or technical reason leaving 299 subjects included in the analysis.
Pre-assignment Details: A total of 304 subjects were enrolled in this study, however, 5 subjects did not receive contrast media due to administrative and /or technical reason leaving 299 subjects included in the analysis.
Groups:
- Arm 1-Iodixanol: Subjects were injected with Iodixanol (Visipaque).
- Arm 2-Iopamidol: Subjects were injected with Iopamidol (Isovue).
Period: Overall Study
Arm/Group | Arm 1-Iodixanol | Arm 2-Iopamidol
Started | 151 | 148
Completed | 148 | 144
Not Completed | 3 | 4
Not completed — Patient received no contrast media | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1-Iodixanol | Arm 2-Iopamidol | Total
Number analyzed (Participants) | 151 | 148 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 91 | 182
  >=65 years | 60 | 57 | 117
Age Continuous [Mean (Standard Deviation); unit: years] | 57.8 (15.23) | 58.5 (15.02) | 58.1 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 80 | 148
  Male | 83 | 68 | 151
Region of Enrollment [Number; unit: participants]
  United States | 65 | 62 | 127
  Germany | 45 | 43 | 88
  Spain | 35 | 35 | 70
  United Kingdom | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Subjects With Moderate/Severe Discomfort When Undergoing Contrast-Enhanced Computed Tomographic (CECT) Imaging of the Abdomen/Pelvis.
Description: Number of subjects experiencing any moderate (score of 4 - 7) to severe (score 8 - 10) discomfort for cold or heat or pain between Iodixanol and Iopamidol.
Time Frame: Within 10 minutes post contrast administration
Measure: Number; unit: Number of Subjects with discomfort
Groups:
- Arm 1-Iodixanol (Visipaque): Subjects injected with Visipaque contrast media. Number of subjects with any Moderate / Severe discomfort.
- Arm 2-Iopamidol (Isovue): Subjects injected with Isovue contrast media. Number of subjects with any Moderate / Severe discomfort.
Arm/Group | Arm 1-Iodixanol (Visipaque) | Arm 2-Iopamidol (Isovue)
Number analyzed (Participants) | 151 | 147
Number of Subjects with discomfort | 53 [27.49 to 42.71] | 99 [59.77 to 74.93]

2. Primary Outcome: Frequency of Subjects With Moderate / Severe Discomfort When Undergoing Contrast-Enhanced Computed Tomographic (CECT) Imaging of the Abdomen/Pelvis.
Description: Number of subjects experiencing moderate (score of 4 -7) to severe (score of 8 - 10) discomfort for cold, heat or pain between Iodixanol and Iopamidol.
Time Frame: Within 10 minutes post contrast administration.
Measure: Number; unit: Number of Subjects with discomfort
Groups:
- Arm 1-Iodixanol (Visipaque 320mgI/mL): Subjects injected with Visipaque 320mgI/mL contrast media. Number of subjects with any Moderate / Severe discomfort.
- Arm 2-Iopamidol (Isovue 370mgI/mL): Subjects injected with Isovue 370mgI/mL contrast media. Number of subjects with any Moderate / Severe discomfort.
Arm/Group | Arm 1-Iodixanol (Visipaque 320mgI/mL) | Arm 2-Iopamidol (Isovue 370mgI/mL)
Number analyzed (Participants) | 151 | 147
Number of Subjects with discomfort
  Discomfort of Cold | 5 [0.46 to 6.17] | 11 [3.23 to 11.74]
  Discomfort of Heat | 45 [22.51 to 37.10] | 94 [56.18 to 71.71]
  Discomfort of Pain | 5 [0.46 to 6.17] | 3 [0.00 to 4.33]

3. Secondary Outcome: Comparison of Overall Image Quality Between Iodixanol and Iopamidol in Patients Undergoing Contrast-Enhanced Computed Tomographic (CECT) Imaging of the Abdomen/Pelvis.
Description: Overall Image Quality rated as 'Excellent, Adequate or Poor' by radiologists blinded to the contrast administration.
Time Frame: Ten minutes post contrast administration.
Measure: Number; unit: Number of subject images
Groups:
- Arm 1-Iodixanol (Visipaque 320mgI/mL): Subjects injected with Visipaque 320mgI/mL contrast media.
- Arm 2-Iopamidol (Isovue 370mgI/mL): Subject injected with Isovue 370mgI/mL contrast media.
Arm/Group | Arm 1-Iodixanol (Visipaque 320mgI/mL) | Arm 2-Iopamidol (Isovue 370mgI/mL)
Number analyzed (Participants) | 151 | 148
Number of subject images
  Image Quality was Excellent | 144 | 133
  Image Quality was Adequate | 7 | 14
  Image Quality was Poor | 0 | 1

ADVERSE EVENTS:
Arm/Group | Arm 1-Iodixanol (Visipaque 320mgI/mL) | Arm 2-Iopamidol (Isovue 370mgI/mL)
Serious Adverse Events (participants affected / at risk) | 0/151 | 1/148
Other Adverse Events (participants affected / at risk) | 121/151 | 134/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Iodixanol (Visipaque 320mgI/mL) (N=151) | Arm 2-Iopamidol (Isovue 370mgI/mL) (N=148)
Acute Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Iodixanol (Visipaque 320mgI/mL) (N=151) | Arm 2-Iopamidol (Isovue 370mgI/mL) (N=148)
Gastrointestinal (Gastrointestinal disorders) | 10 (10) | 10 (10)
General disorder: Feeling Cold (General disorders) | 8 (8) | 8 (8)
Nervousness (Nervous system disorders) | 13 (13) | 9 (9)
General Disorders: Feeling Hot (General disorders) | 77 (77) | 92 (92)
Administration Site Conditions: Injection Site Coldness (General disorders) | 5 (5) | 9 (9)
Administration Site Conditions: Injection Site Reaction (General disorders) | 30 (30) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No